CLINICAL TRIAL: NCT06040047
Title: Identifying Patients With Cervical Radiculopathy Responding to Proprioceptive Neuromuscular Facilitation Exercises Combined With Passive Cervical Mobilization: Clinical Prediction Rule
Brief Title: Prediction of Cervical Radiculopathy Success With PNF and Mobilization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed ElMelhat, lecturer, orthopedic physiotherapy department, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 012/002739
Record Dates: First submitted 2023-09-10; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Cervical Radiculopathy
MeSH Terms: conditions — Radiculopathy | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PNF plus mobilization (Experimental): This single group will receive passive mobilization and proprioceptive neuromuscular facilitation for cervical region.
  Interventions: Other: Proprioceptive neuromuscular facilitation; Other: Passive mobilization

INTERVENTIONS:
Other: Proprioceptive neuromuscular facilitation — Contract relax technique for each neck motion for three repetitions.
  Other Names: PNF
Other: Passive mobilization — To restore normal joint play, postero-anterior passive joint mobilization of cervical spine segments and cervicothoracic junction in limited motion will be applied.

SUMMARY:
The goal of this predictive interventional study is todetrmine clinical predictors for success with combined proprioceptive neuromusclualr faciitaion (PNF) and passive mobilization ain patients with cervical radiculopathy (CR).

DETAILED DESCRIPTION:
This study will answer the question, what are the factors affecting success with PNF and mobilization for patients with CR? No control group. The goal of this new study is to see the effect of age, duration of symptoms, forward posture angle and neck disability index response to passive mobilization combined with the PNF technique

ELIGIBILITY:
Inclusion Criteria:

* Participants with cervical radiculopathy.
* Age ranges between 40 and 60 years old.
* Minimum score (3 out of 10-point) on a visual analog scale (VAS)
* Orthopedic clinical confirmation reveals a history of neck pain.

Exclusion Criteria:

* Whiplash injury.
* Previous Cervical surgery.
* Pain less than three months.
* Mechanical and non-specific neck pain.
* Pregnancy.
* Bilateral arm pain.
* Inflammatory arthritides.
* Osteoporosis.
* Symptoms of vertebrobasilar insufficiency.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Cervical pain | 6 weeks
  Score on numeric pain rating scale (points)
Cervical disability | 6 weeks
  Disability will be measured with Northwick Park neck pain Questionnaire.

SECONDARY OUTCOMES:
Cervical proprioception | 6 weeks
  Cervical joint position error will be measured with laser pointer.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed ElMelhat, Phd, Principal Investigator — Cairo University
Locations (1):
- ME, Cairo, Egypt